CLINICAL TRIAL: NCT02025010
Title: Phase II Clinical Trial of Abiraterone Acetate Without Exogenous Glucocorticoids in Men With Castration-resistant Prostate Cancer With Correlative Assessment of Hormone Intermediates.
Brief Title: Study of Abiraterone Acetate Without Exogenous Glucocorticoids in Men With Castration-resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Principal Investigator, Mary-Ellen Taplin, MD, Principal Investigators, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-449
Record Dates: First submitted 2013-12-13; First posted 2013-12-31 (Estimated); Results first posted 2022-11-08 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Castration-resistant Prostate Cancer
Keywords: Castration-resistant Prostate Cancer; Abiraterone Acetate
MeSH Terms: interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- abiraterone acetate (Experimental): Participants will be treated with four 250 mg tablets (1,000 mg) of abiraterone acetate (AA) orally on 28-day cycles. For participants who experience persistent or severe mineralocorticoid excess or have PSA progression, prednisone 5 mg by mouth twice daily will be added.
  Patients will be treated until radiographic disease progression and unacceptable AE or taken off study for other reason.
  Interventions: Drug: abiraterone acetate

INTERVENTIONS:
Drug: abiraterone acetate — Abiraterone acetate is a selective and irreversible inhibitor of CYP17 which has demonstrated clinical efficacy in patients with CRPC. Currently, AA is administered with concomitant prednisone.
  Other Names: JNJ21208

SUMMARY:
This study is comparing the safety and effectiveness of abiraterone acetate alone, followed by the addition of prednisone (when the participant's disease worsens or the physician feels it would lessen symptoms of toxicity) versus the current approved treatment regimen which involves the concomitant use of prednisone in conjunction with abiraterone acetate. Additionally, this study is also examining why participants stop responding to treatment with abiraterone acetate by evaluating blood and tissue.

DETAILED DESCRIPTION:
Participants will be treated with abiraterone acetate (AA) in 28-day cycles. Participants will be monitored (weekly for the first two cycles, then on Day 1 of each subsequent cycle) for symptoms of persistent or severe mineralocorticoid excess (including hypertension, hypokalemia).

For participants who experience symptoms of persistent or severe hypertension or hypokalemia as detailed in the above schema, prednisone 5 mg by mouth twice daily will be added. We will monitor for other symptoms of AA toxicity to include fluid retention and fatigue.

For participations who tolerate AA monotherapy without the addition of prednisone to manage symptoms of persistent or severe mineralocorticoid excess, prednisone 5 mg by mouth twice daily will be added at Prostate Specific Antigen (PSA) progression. Participants will be continued on study until symptomatic or radiographic progression or taken off study for another reason as detailed in protocol.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* Be a male ≥ 18 years of age.
* Participants must have histologically or cytologically confirmed adenocarcinoma of the prostate without >50% neuroendocrine differentiation or small cell histology.
* Participants must have progressive disease as defined by one or more of the following:
* Castrate resistant disease as defined by Prostate cancer working Group (PCWG).[30] Participants must have a rise in PSA on two successive determinations at least one week apart and PSA levels ≥ 2 ng/ml (only the screening PSA needs to be ≥ 2 ng/ml) and testosterone levels < 50 ng/dL.
* Soft tissue progression defined by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
* Bone disease progression defined by Prostate Cancer Clinical Trials Working Group 2 (PCWG2) with two or more new lesions on bone scan.[30]
* Castration-resistant prostate cancer (CRPC) with metastatic disease with at least one site of metastatic disease must be amenable to needle biopsy. Soft tissue biopsy sites include: lymph node or visceral metastases. Bone sites include lumbar vertebrae, pelvic bones and long bones. Excluded sites are thoracic, cervical vertebrae, skull and rib lesions. Biopsy site will be selected with guidance of interventional radiologist determining best site to optimize balance of obtaining useful tissue for analysis and minimizing risk.
* Participants without orchiectomy must be maintained on Luteinizing hormone-releasing hormone (LHRH) agonist/antagonist therapy.
* Participants may have had any number of previous hormonal therapies (antiandrogens including enzalutamide, steroids, estrogens, finasteride, dutasteride, ketoconazole) provided these were discontinued ≥ 4 weeks before starting the trial.
* Participants may have had up to two previous cytotoxic therapeutic regimens provided these were discontinued ≥ 4 weeks before starting the trial.
* At least a 4 week interval from previous prostate cancer treatment other than LHRH agonist/antagonist therapy or bisphosphonates to the start of protocol therapy.
* Participants receiving bisphosphonates therapy can be maintained on this therapy. If participants have not started bisphosphonates, it is recommended that they start treatment after the first biopsy.
* Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Karnofsky >60%, see Appendix A).

Participants must have normal organ and marrow function as defined below:

* Platelets > 50,000/microliter (mcL)
* Serum potassium ≥ 3.5 mmol/L (independent of potassium supplementation)
* Serum albumin ≥ 3.0 g/dL
* Aspartate transaminase (AST), Alanine transaminase (ALT), and total bilirubin ≤ 1.5 x Institutional Upper Limit of Normal (ULN).
* Partial thromboplastin time (PTT) ≤ 60, International Normalized Ratio (INR) ≤ 1.5 Institutional ULN unless on warfarin therapy (investigator would need to determine if safe for participant to stop warfarin prior to biopsy)
* Controlled blood pressure (systolic blood pressure < 140 and diastolic blood pressure <90) on no more than three anti-hypertensive agents. Drug formulations containing two or more anti-hypertensive agents will be counted based on the number of active agents in each formulation.
* EKG showing a normal QTc interval (QTc < 450 msec).
* Left ventricular ejection fraction ≥ 50%.
* Have signed an informed consent document indicating that the subjects understands the purpose of and procedures required for the study and are willing to participate in the study.
* Be willing/able to adhere to the prohibitions and restrictions specified in this protocol.
* Written Authorization for Use and Release of Health and Research Study Information (US sites only) has been obtained.
* Able to swallow the study drug whole as a tablet.
* Willing to take AA on an empty stomach; no food should be consumed at least two hours before and for at least one hour after the dose AA is taken.
* Participants who have partners of childbearing potential must be willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the PI during the treatment period and for 1 week after last dose of AA.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Uncontrolled illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or would make prednisone/prednisolone (corticosteroid) use contraindicated.
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class III or IV heart disease or cardiac ejection fraction measurement of < 50 % at baseline.
* Thromboembolism within 6 months of Cycle 1, Day 1.
* Severe hepatic impairment (Child-Pugh Class C).
* History of pituitary or adrenal dysfunction.
* Poorly controlled diabetes.
* History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug.
* Have a pre-existing condition that warrants long-term corticosteroid use.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: 1) individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy, or 2) individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: superficial bladder cancer, basal cell or squamous cell carcinoma of the skin.
* Known brain metastasis.
* Prior therapy with AA.
* Have known allergies, hypersensitivity, or intolerance to AA or prednisone or their excipients.
* Surgery or local prostatic intervention within 30 days of the first dose. In addition, any clinically relevant issues from the surgery must have resolved prior to Cycle 1, Day 1.
* Major surgery or radiation therapy within 4 weeks of Cycle 1, Day 1.
* Strontium-89 or samarium-153 therapy within 4 weeks of Cycle 1, Day 1.
* Radiotherapy, chemotherapy or immunotherapy within 4 weeks, or single fraction of palliative radiotherapy within 14 days of administration of Cycle 1, Day 1.
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of Cycle 1, Day 1.
* Any acute toxicities due to prior chemotherapy and/or radiotherapy that have not resolved to a NCI Common Toxicity Criteria for Adverse Effects (CTCAE) version 4 grade of ≤ 1. Chemotherapy induced alopecia and grade 2 peripheral neuropathy are allowed.
* Condition or situation which, in the investigator's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with participant's participation in the study.
* Individuals not willing to comply with the procedural requirements of this protocol.
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AA.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01-27 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2025-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ellen Taplin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center West Harrison, Harrison, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center Sleepy Hollow, Sleepy Hollow, New York

REFERENCES:
- [Derived] Sperger JM, Emamekhoo H, McKay RR, Stahlfeld CN, Singh A, Chen XE, Kwak L, Gilsdorf CS, Wolfe SK, Wei XX, Silver R, Zhang Z, Morris MJ, Bubley G, Feng FY, Scher HI, Rathkopf D, Dehm SM, Choueiri TK, Halabi S, Armstrong AJ, Wyatt AW, Taplin ME, Zhao SG, Lang JM. Prospective Evaluation of Clinical Outcomes Using a Multiplex Liquid Biopsy Targeting Diverse Resistance Mechanisms in Metastatic Prostate Cancer. J Clin Oncol. 2021 Sep 10;39(26):2926-2937. doi: 10.1200/JCO.21.00169. Epub 2021 Jul 1. PMID 34197212

RESULTS

PARTICIPANT FLOW:
Groups:
- Abiraterone Acetate: Participants will be treated with four 250 mg tablets (1,000 mg) of abiraterone acetate (AA) orally on 28 day cycles. For participants who experience symptoms of persistent or severe mineralocorticoid excess or PSA progression, prednisone 5 mg by mouth twice daily will be added.
Period: Overall Study
Arm/Group | Abiraterone Acetate
Started | 60
Completed | 0
Not Completed | 60
Not completed — Symptomatic or radiographic progression | 36
Not completed — Adverse Event | 6
Not completed — Physician Decision | 7
Not completed — Withdrawal by Subject | 3
Not completed — Intercurrent illness | 3
Not completed — Patients still on treatment | 3
Not completed — Never initiate the treatment | 2

BASELINE CHARACTERISTICS:
Population: Patients who received at least 1 dose of abiraterone acetate
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 58
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [61 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 53
  More than one race | 0
  Unknown or Not Reported | 3
Baseline antihypertensive use [Count of Participants; unit: Participants]
  Any | 26
  1 agent | 15
  2 agents | 8
  3 agents | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Toxicities That Required the Addition of Prednisone to Manage Symptoms of Persistent or Severe Mineralocorticoid Excess
Description: Patients requiring prednisone to manage toxicities such as COU-302 any grade or COU-301 grade 3-4 hypertension, hypokalemia and edema per CTCAE v. 4.0 were summarized using frequency and percentage.
Time Frame: Patients were on abiraterone acetate up to 57 months and toxicities of mineralocorticoid excess were monitored each cycle (1cycle = 28 days).
Population: Participants who received at least 1 dose of abiraterone acetate.
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 58
Participants
  Any grade mineralocorticoid toxicities | 38
  Any grade hypertension | 28
  Any grade hypokalemia | 15
  Any grade edema | 11
  Grade 3-4 mineralocorticoid toxicities | 12
  Grade 3-4 hypertension | 9
  Grade 3-4 hypokalemia | 4
  Grade 3-4 edema | 0

2. Secondary Outcome: Safety and Tolerability Associated With AA Monotherapy and the Addition of Prednisone to AA.
Description: Grade 3 or higher toxicities attribution to AA monotherapy with or without prednisone were summarized descriptively.
Time Frame: Adverse events were assessed continuously on treatment and up to 30 days after going off treatment (up to 55 months).
Population: Patients who initiated at least one dose of abiraterone acetate. Prednisone was co-administered for 35 patients who experienced symptoms of persistent or severe mineralocorticoid excess or PSA progression at any cycle.
Measure: Count of Participants; unit: Participants
Groups:
- Abiraterone Acetate: Participants will be treated with abiraterone acetate (AA) in 28-day cycles. Participants will be monitored (weekly for the first two cycles, then on Day 1 of each subsequent cycle) for symptoms of persistent or severe mineralocorticoid excess (including hypertension, hypokalemia). For participants who experience symptoms of persistent or severe hypertension or hypokalemia as detailed in the above schema, prednisone 5 mg by mouth twice daily will be added.
- Abiraterone Acetate + Prednisone: Prednisone 5mg by mouth twice was co-administered with abiraterone acetate for those who experience symptoms of persistent or severe mineralocorticoid excess or PSA progression at any cycle. This is subset of the patients who initiated abiraterone acetate (n=58).
Arm/Group | Abiraterone Acetate | Abiraterone Acetate + Prednisone
Number analyzed (Participants) | 58 | 35
Participants
  Grade 3 Anemia | 0 | 1
  Grade 3 Depression | 0 | 1
  Grade 3 Hypertension | 9 | 2
  Grade 3 Hypokalemia | 2 | 2
  Grade 3 Mood Alteration | 0 | 1
  Grade 4 Hypertension | 0 | 1
  Grade 3 Alanine aminotransferase increased | 1 | 0
  Grade 3 Aspartate aminotransferase increased | 1 | 0
  Grade 3 Fatigue | 1 | 0
  Grade 3 Gastrointestinal Bleed | 1 | 0
  Grade 3 Rash pustular | 1 | 0
  AE grade <3 | 40 | 27
  No AE reported post baseline | 2 | 0

3. Secondary Outcome: Number of Participants Requiring the Addition of Prednisone to Manage Symptoms of Severe Fatigue.
Description: Participants initiated treatment with prednisone for ≥grade 3 fatigue were summarized using frequency and percentage.
Time Frame: Patients were on abiraterone acetate up to 57 months.
Population: Patients receiving at least 1 dose of abiraterone acetate.
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 58
Participants | 1

4. Secondary Outcome: Changes in Serum Concentrations of Corticosteroid Intermediates Between the First and Second Assessment Visits.
Description: Percent change in corticosterone level between the first visit and the second visit was summarized by whether patients initiated prednisone for hypertension and hypokalemia.
Time Frame: 1 month
Population: Patients who received at least one dose of abiraterone acetate and had available serum concentrations of corticosteroid.
Measure: Median (Inter-Quartile Range); unit: Percentage
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 56
Percentage
  Patients without prednisone: number analyzed (Participants) | 49
  Patients without prednisone | 58 [30 to 93]
  Patients with prednisone: number analyzed (Participants) | 7
  Patients with prednisone | 116 [30 to 248]

5. Secondary Outcome: Changes in Serum Concentrations of ACTH Between Cycle 1 and Cycle 2.
Description: Changes in serum concentrations of ACTH at second assessment referent to the value at the first visit were summarized descriptively.
Time Frame: 1 month
Population: Patients receiving at least one dose of abiraterone acetate
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 58
pg/mL | 0 [0 to 49.5]

6. Secondary Outcome: Percent Changes in Serum Concentrations of Androgen (Including Testosterone, DHT and Androgen Precursors) Between Cycle 1 and Cycle 2.
Description: Change in corticosterone level between cycle 2 and cycle 1 was summarized by whether patients initiated prednisone for hypertension and hypokalemia.
Time Frame: 1 month
Population: Patients who initiated abiraterone acetate (n=58) and had available each serum hormone data at cycles 1 and 2 (can be smaller than 58).
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 58
Percent change
  Androstenedione change among patients without prednisone: number analyzed (Participants) | 19
  Androstenedione change among patients without prednisone | -0.97 [-0.99 to -0.94]
  Androstenedione change among patients with prednisone: number analyzed (Participants) | 21
  Androstenedione change among patients with prednisone | -0.97 [-0.98 to -0.94]
  Androsterone change among patients without prednisone: number analyzed (Participants) | 19
  Androsterone change among patients without prednisone | -0.91 [-0.95 to -0.82]
  Androsterone change among patients with prednisone: number analyzed (Participants) | 21
  Androsterone change among patients with prednisone | -0.87 [-0.93 to -0.79]
  Corticosterone change among patients without prednisone: number analyzed (Participants) | 19
  Corticosterone change among patients without prednisone | 42.7 [16.9 to 93.4]
  Corticosterone change among patients with prednisone: number analyzed (Participants) | 21
  Corticosterone change among patients with prednisone | 51.7 [34.3 to 96.4]
  Cortisol change among patients without prednisone: number analyzed (Participants) | 19
  Cortisol change among patients without prednisone | -0.58 [-0.81 to -0.46]
  Cortisol change among patients with prednisone: number analyzed (Participants) | 21
  Cortisol change among patients with prednisone | -0.73 [-0.79 to -0.66]
  DHEA change among patients without prednisone: number analyzed (Participants) | 19
  DHEA change among patients without prednisone | -0.98 [-0.99 to -0.95]
  DHEA change among patients with prednisone: number analyzed (Participants) | 21
  DHEA change among patients with prednisone | -0.99 [-0.99 to -0.97]
  DHT change among patients without prednisone: number analyzed (Participants) | 19
  DHT change among patients without prednisone | -0.37 [-0.52 to 0]
  DHT change among patients with prednisone: number analyzed (Participants) | 21
  DHT change among patients with prednisone | -0.29 [-0.47 to 0]
  11 Deoxycorticosterone change among patients without prednisone: number analyzed (Participants) | 18
  11 Deoxycorticosterone change among patients without prednisone | 40.3 [21.7 to 83.2]
  11 Deoxycorticosterone change among patients with prednisone: number analyzed (Participants) | 21
  11 Deoxycorticosterone change among patients with prednisone | 47.8 [33.0 to 77.5]
  11 Deoxycortisol change among patients without prednisone: number analyzed (Participants) | 18
  11 Deoxycortisol change among patients without prednisone | -0.61 [-0.79 to -0.43]
  11 Deoxycortisol % change among patients with prednisone: number analyzed (Participants) | 21
  11 Deoxycortisol % change among patients with prednisone | -0.71 [-0.86 to -0.64]
  17 Hydroxypregnenolone % change among patients without prednisone: number analyzed (Participants) | 19
  17 Hydroxypregnenolone % change among patients without prednisone | 0 [-0.12 to 1.23]
  17 Hydroxypregnenolone % change among patients with prednisone: number analyzed (Participants) | 21
  17 Hydroxypregnenolone % change among patients with prednisone | 0 [-0.19 to 0.59]
  17 Hydroxyprogesterone change among patients without prednisone: number analyzed (Participants) | 19
  17 Hydroxyprogesterone change among patients without prednisone | 0.02 [-0.41 to 0.92]
  17 Hydroxyprogesterone change among patients with prednisone: number analyzed (Participants) | 21
  17 Hydroxyprogesterone change among patients with prednisone | 0.06 [-0.32 to 0.67]
  Pregnenolone change among patients without prednisone: number analyzed (Participants) | 18
  Pregnenolone change among patients without prednisone | 19.0 [15.5 to 25.8]
  Pregnenolone change among patients with prednisone: number analyzed (Participants) | 21
  Pregnenolone change among patients with prednisone | 23.4 [18.9 to 31.4]
  Progesterone change among patients without prednisone: number analyzed (Participants) | 19
  Progesterone change among patients without prednisone | 96.3 [31.0 to 132.5]
  Progesterone change among patients with prednisone: number analyzed (Participants) | 21
  Progesterone change among patients with prednisone | 104.6 [63.7 to 201.5]
  Testosterone change among patients without prednisone: number analyzed (Participants) | 51
  Testosterone change among patients without prednisone | 0.07 [0.04 to 0.1]
  Testosterone change among patients with prednisone: number analyzed (Participants) | 7
  Testosterone change among patients with prednisone | 0.07 [0.06 to 0.08]

7. Secondary Outcome: Changes in BMI Between Cycle 1 and Next Cycle
Description: Changes in BMI between cycle 1 and cycle 2 were summarized descriptively.
Time Frame: 1 month
Population: Patients receiving at least one dose of abiraterone acetate.
Measure: Median (Inter-Quartile Range); unit: kg/m²
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 58
kg/m² | 0 [0 to 0.15]

8. Secondary Outcome: Changes in Hemoglobin-A1c Between Cycle 1 and Next Cycle (Cycle 4)
Description: Changes in HbA1c at cycle 1 and next measurement at cycle 4 were summarized descriptively.
Time Frame: 3 months
Population: Patients receiving at least one dose of abiraterone acetate.
Measure: Median (Inter-Quartile Range); unit: Percentage of glycated hemoglobin
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 58
Percentage of glycated hemoglobin | 0 [-0.2 to 0]

9. Secondary Outcome: PSA Response and Its Duration to AA Monotherapy.
Description: PSA response was defined per PCWG2 criteria (PSA reduction of ≥50%) and duration of PSA response is defined as time from PSA response to PSA progression or death, whichever occurs first.
Time Frame: PSA was measured every cycle (up to 25 months)
Population: PSA responders after receiving at least one dose of abiraterone acetate without prednisone
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 22
months | 3 [1 to 18]

10. Secondary Outcome: PSA Response and Its Duration to Addition of Prednisone to AA at Time of PSA Progression on AA Monotherapy.
Description: Among those who initiated prednisone due to PSA progression, duration of PSA response was calculated as time from PSA response (PSA reduction ≥50%) to PSA progression or death, whichever occurs first.
Time Frame: PSA was measured every cycle (up to 25 months)
Population: Patients who achieved a PSA response and initiated prednisone at PSA progression
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 22
months | 5 [2 to 8]

11. Secondary Outcome: Response of Measurable Disease to AA Monotherapy.
Description: Radiographic response of measurable disease is defined using RECIST v 1.1 for soft-tissue and visceral disease and PCWG2 for bone disease.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Response is tabulated descriptively.
Time Frame: Imaging was performed every 12 weeks up to 23 months.
Population: Patients who received at least 1 dose of abiraterone acetate without prednisone and had a measurable disease at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 11
Participants
  Complete response | 1
  Partial response | 2
  Stable disease | 4
  Progressive disease | 4

12. Secondary Outcome: Number of Patients Who Received AA Monotherapy and Progressed With Measurable Disease at Pre-study
Description: Radiographic disease progression is defined using RECIST v 1.1 for soft-tissue and visceral disease and PCWG2 for bone disease (2 or more new lesions on bone scan and for the first 12-week assessment, defining disease progression requires a confirmatory scan performed 6 or more weeks later which shows a minimum of 2 additional new lesions).
Time Frame: Imaging was performed every 12 weeks up to 23 months.
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 11
Participants | 5

13. Secondary Outcome: Response of Measurable Disease to Addition of Prednisone to AA at Time of PSA Progression on AA Monotherapy.
Description: as for outcome 11
Time Frame: Imaging was performed every 12 weeks up to 23 months.
Population: Patients who received at least one dose of abiraterone acetate with prednisone at PSA progression and had a measurable disease at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 10
Participants
  Complete response | 3
  Partial response | 1
  Stable disease | 5
  Progressive disease | 1

14. Secondary Outcome: Number of Patients Who Progressed With Measurable Disease at Pre-study Among Those Who Were Added of Prednisone to AA at Time of PSA Progression on AA Monotherapy.
Description: Radiographic response of measurable disease is defined using RECIST v 1.1 for soft-tissue and visceral disease and PCWG2 for bone disease. Due to small number patients, patients who experienced progressive disease were summarized using frequency and time to progression using Kaplan-Meier method was not calculated.
Time Frame: Imaging was performed every 12 weeks up to 23 months.
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 10
Participants | 6

15. Secondary Outcome: Subsequent Lines of Therapy
Description: Subsequent lines of therapy following study drug discontinuation were not collected for this trial.
Time Frame: Data not collected.
Population: Data not collected.
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Toxicities were assessed every cycle and up to 30 days after coming off treatment. Toxicities were collected up to around 55 months.
Description: A serious adverse event (SAE) is any adverse event, occurring at any dose and regardless of causality that:
  Results in death Is life-threatening. Life-threatening means that the person was at immediate risk of death from the reaction as it occurred, i.e., it does not include a reaction which hypothetically might have caused death had it occurred in a more severe form.
  Requires or prolongs inpatient hospitalization Results in persistent or significant disability/incapacity
Arm/Group | Abiraterone Acetate
All-Cause Mortality (participants affected / at risk) | 24/60
Serious Adverse Events (participants affected / at risk) | 9/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate (N=60)
Anemia (Blood and lymphatic system disorders) | 1
Heart failure (Cardiac disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Lung infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Creatinine increased (Investigations) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate (N=60)
Anemia (Blood and lymphatic system disorders) | 4
Chest pain - cardiac (Cardiac disorders) | 2
Heart failure (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 2
Sinus bradycardia (Cardiac disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 4
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 3
Vertigo (Ear and labyrinth disorders) | 2
Blurred vision (Eye disorders) | 2
Optic nerve disorder (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 8
Stomach pain (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4
Chills (General disorders) | 1
Edema limbs (General disorders) | 11
Edema trunk (General disorders) | 1
Fatigue (General disorders) | 45
Fever (General disorders) | 1
Gait disturbance (General disorders) | 1
Localized edema (General disorders) | 2
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 22
General disorders and administration site conditions - Other, specify (General disorders) | 2
Papulopustular rash (Infections and infestations) | 1
Prostate infection (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 2
Wound infection (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 4
Bruising (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 6
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 12
Blood bilirubin increased (Investigations) | 2
Creatinine increased (Investigations) | 2
Lipase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1
Serum amylase increased (Investigations) | 1
Weight gain (Investigations) | 3
Weight loss (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 21
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 5
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 7
Paresthesia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 7
Syncope (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 2
Restlessness (Psychiatric disorders) | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 3
Hematuria (Renal and urinary disorders) | 3
Renal calculi (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 15
Urinary incontinence (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 3
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 7
Erectile dysfunction (Reproductive system and breast disorders) | 1
Gynecomastia (Reproductive system and breast disorders) | 3
Pelvic pain (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Skin atrophy (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2
Hot flashes (Vascular disorders) | 26
Hypertension (Vascular disorders) | 31
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT02025010/Prot_SAP_000.pdf